CLINICAL TRIAL: NCT01536691
Title: To Assess the Efficacy and Safety of Ramosetron, Aprepitant and Dexamethasone Therapy vs Ondansetron, Aprepitant and Dexamethasone Therapy for Preventing of Nausea and Vomiting in Highly Emetogenic Chemotherapy (ROAD Study)
Brief Title: Ramosetron, Aprepitant and Dexamethasone Versus Ondansetron, Aprepitant and Dexamethasone
Acronym: ROAD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hallym University Medical Center (Other)
Collaborators: Korean Cancer Study Group (Other); Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ROAD
Record Dates: First submitted 2011-10-04; First posted 2012-02-22 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-02

CONDITIONS: Cancer; Malignancy
Keywords: ramosetron; ondansetron; aprepitant; chemotherapy induced nausea & vomiting
MeSH Terms: conditions — Neoplasms; Vomiting | interventions — ramosetron; Ondansetron

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ramosetron, aprepitant, dexamethasone (Experimental): ramosetron 0.3 mg iv D1 aprepitant 125 mg po D1, 80 mg po D2, 80 mg po D3 dexamethasone 12 mg po D1, 8 mg po D2-4
  Interventions: Drug: ramosetron
- ondansetron, aprepitant, dexamethasone (Active Comparator): ondansetron 16 mg iv D1 aprepitant 125 mg po D1, 80 mg po D2, 80 mg po D3 dexamethasone 12 mg po D1, 8 mg po D2-4
  Interventions: Drug: ondansetron

INTERVENTIONS:
Drug: ramosetron — ramosetron 0.3 mg iv D1 aprepitant 125 mg po D1, 80 mg po D2, 80 mg po D3 dexamethasone 12 mg po D1, 8 mg po D2-4
  Other Names: Nasea - ramosetron; Emend - aprepitant
  Arms: ramosetron, aprepitant, dexamethasone
Drug: ondansetron — ondansetron 16 mg iv D1 aprepitant 125 mg po D1, 80 mg po D2, 80 mg po D3 dexamethasone 12 mg po D1, 8 mg po D2-4
  Other Names: zofran - ondansetron; Emend - aprepitant
  Arms: ondansetron, aprepitant, dexamethasone

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Ramosetron, Aprepitant and Dexamethasone therapy versus Ondansetron, Aprepitant and Dexamethasone therapy for preventing of nausea and vomiting in highly emetogenic chemotherapy (ROAD study):

Prospective multicenter, randomized, single blinded, phase III study.

DETAILED DESCRIPTION:
To assess the efficacy and safety of Ramosetron, Aprepitant and Dexamethasone therapy versus Ondansetron, Aprepitant and Dexamethasone therapy for preventing of nausea and vomiting in highly emetogenic chemotherapy (ROAD study):

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as malignancy who will be treated with highly emetogenic chemotherapeutic agents (NCCN guideline v1.0 2011 anti-emesis), over 20 years and both sex
2. ECOG performance status 0-2
3. Available oral administration of study drugs
4. Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policy of the hospital

Exclusion Criteria:

1. Severe Hypertension, severe Heart disease, kidney disease (serum creatinine > 3 mg/dl), liver disease (AST, ALT > 3 times of upper normal range, ALP > 2 times of upper normal range)
2. Patients with GI obstruction, active gastric ulcer or other diseases that could provoke nausea and vomiting
3. Patients who have nausea and vomiting within 1 week before chemotherapy
4. Patients who should take steroid, antiemetics, pimozide, terfenadine, astemizole, cisapride, rifampin, carbamazepine, phenytoin, ketoconazole, itraconazole, nefazodone, troleandomycin, clarithromycin, ritonavir or nelfinavir for the treatment of other diseases
5. Patients with brain tumor, brain metastasis or seizure
6. Patients receiving chemotherapy within 12 months before enrollment
7. Patients who need radiation therapy during study period or receiving radiation therapy within 2 weeks before chemotherapy
8. Patients who have known allergy or severe side effect on study drugs
9. Pregnant or lactating women, or women who wish to become pregnant
10. Others whom the investigator judges inappropriate as subjects for this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-11 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
complete response (CR) | acute phase (within 24 hrs after onset of chemotherapy)
  CR means no vomiting & no rescue medication

SECONDARY OUTCOMES:
complete response | during delayed phase and whole study period
  Delayed phase means 'from day 2 to day 5' after onset of chemotherapty whole study period means 'from day 1 to day 5' after onset of chemotherapty (acute phase + delayed phase).

CONTACTS AND LOCATIONS:
Overall Officials: Sangwon Shin, M.D., Principal Investigator — Korea University Anam Hospital
Locations (1):
- Hyo Jung Kim, Anyang-si, Gyeonggi-do, South Korea